CLINICAL TRIAL: NCT00260780
Title: The MISTERS Project: An STD Prevention Intervention for Men Newly Released From Jail
Brief Title: An STD Prevention Intervention for Men Newly Released From Jail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: STAND, Inc. (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3728; U52/CCU422491; H25/CCH404332-11
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2005-12-02 (Estimated); Status verified 2005-12

CONDITIONS: Sexually Transmitted Diseases; Risk Behavior
Keywords: sexually transmitted diseases; Risk Behavior
MeSH Terms: conditions — Sexually Transmitted Diseases; Risk-Taking

INTERVENTIONS:
Behavioral: The MISTERS Intervention for Post Jail Release Men

SUMMARY:
Study participants who are exposed to the intervention will: 1)report more condom use during sexual episodes; 2) have fewer new and repeat STD infections 3)demonstrate greater risk reduction, communication, and anger management skills; 4) report fewer substance use behaviors, and 5)report more health care seeking activities, than the participants in the control group

DETAILED DESCRIPTION:
The MISTERS study is a randomized control trial of a cognitive-behavioral skill building multi-session intervention that targets men who are newly released from jail and have a history of drug use. Men 45 days or less post release with self reported HIV negative and substance use histories were randomized into either a 5-session intervention or control group. Study participation included four time-sensitive interviews and STD testing at three time periods. The interview questions included demographics, STD history and knowledge, sexual risk behaviors, as well as an assessment of anger management, communication, and condom use skills.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 to 60, English speaking, not in jail for sexual offenses (rape or child molestation), reported risk behavior in two months prior to incarceration, weekday and evening availability, viable contact information, self-reported HIV negative status, released from jail no more than 45 days prior, and not visibly under the influence of drugs or alcohol at the time of eligibility determination

Exclusion Criteria:

* Opposite of the above

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300
Dates: Start 2001-06; Study Completion 2004-06

PRIMARY OUTCOMES:
Change in risk behaviors

SECONDARY OUTCOMES:
Reported STDs

CONTACTS AND LOCATIONS:
Overall Officials: Samantha P Williams, Ph.D., Study Chair — CDC/NCHSTP/DSTDP/BIRB; Charles Sperling, M.S., Principal Investigator — STAND, Inc.
Locations (1):
- STAND, Inc., Decatur, Georgia, United States